CLINICAL TRIAL: NCT04477694
Title: The Effect of Diabetes Mellitus on Hemodynamics, Procedure Times, Anesthetic Consumption and Complications in Colonoscopy Under Sedoanalgesia
Brief Title: The Effect of Diabetes Mellitus in Colonoscopy Under Sedoanalgesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Yonca Özvardar Pekcan, MD, Anesthesia and Reanimation specialist, principal Investigator, Baskent University
Other Study IDs: K19/320
Record Dates: First submitted 2020-06-29; First posted 2020-07-20 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus, Type 2; Sedoanalgesia
Keywords: Diabetes mellitus; Sedoanalgesia; Colonoscopy under sedoanalgesia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- type II diabetic patients
  Interventions: Procedure: colonoscopy under sedoanalgesia
- non-diabetic patients
  Interventions: Procedure: colonoscopy under sedoanalgesia

INTERVENTIONS:
Procedure: colonoscopy under sedoanalgesia — Colonoscopy is a widely used method for diagnosing and treating colonic diseasea with a thin, flexible camera.

SUMMARY:
INTRODUCTION AND AIM Diabetes Mellitus (DM) is a common endocrine disease in the world. Colon polyps and colorectal cancers are reported more in DM patients. Therefore diabetic patients are recommended to have colonoscopy frequently. The aim of this study is to search the effect of DM on hemodynamics, procedure times, anesthetic consumption and complications in colonoscopy under sedoanalgesia.

MATERIALS AND METHODS Following Institutional Review Board and Ethics Committee approval of Başkent University, this study is planned to be prospective and double-blind in 50 type II diabetic and 50 non-diabetic ASA I-II, aged between 18-65 years female patients scheduled for elective colonoscopy under sedoanalgesia. Exclusion criteria are age outside the range of 18-65 years, ASA phsical status ≥ 3, inability to provide informed consent, pregnancy, previous adverse reactions to medications used in the study, history of anesthesia and sedation in the last 7 days, psychiatric or emotional disorders, addiction to the opioids or sedatives used in the study, diabetic nephrophathy, high BUN and creatinine values, advanced stages of diabetic nonalcoholic liver disease and high liver function tests, diabetic sensorymotor and autonomic neuropathy.

After sedoanalgesia is applied systolic and diastolic blood pressure, heart rate, SpO2, respiratory rate, RSS, MPADS, procedure times, total anesthetic doses, stomach ache and other effects will be recorded.

EXPECTATIONS AND SCIENTIFIC CONTRIBUTIONS There is evidence about determining the risks that diabetic patients have during colonoscopy and applying a special patient care protocol for these patients is suggested to improve the procedure and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged between 18-65 years old
* Type II diabetic and non-diabetic

Exclusion Criteria:

* Age outside the range of 18-65 years
* ASA phsical status ≥ 3
* Inability to provide informed consent
* Pregnancy
* Previous adverse reactions to medications used in the study
* History of anesthesia and sedation in the last 7 days
* Psychiatric or emotional disorders
* Addiction to the opioids or sedatives used in the study
* Diabetic nephrophathy, high BUN and creatinine values
* Advanced stages of diabetic nonalcoholic liver disease and high liver function tests
* Diabetic sensorymotor and autonomic neuropathy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Type II diabetic and non-diabetic ASA I-II, aged between 18-65 years female patients scheduled for elective colonoscopy under sedoanalgesia
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12-27 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of mean blood pressure in diabetic and non-diabetic patients in colonoscopy under sedoanalgesia | 24 hour
  After sedoanalgesia is applied mean blood pressure will be recorded.
Comparison of heart rate in diabetic and non-diabetic patients in colonoscopy under sedoanalgesia | 24 hour
  After sedoanalgesia is applied heart rate will be recorded.
Comparison of SpO2 in diabetic and non-diabetic patients in colonoscopy under sedoanalgesia | 24 hour
  After sedoanalgesia is applied SpO2 will be recorded.
Comparison of respiratuar rate in diabetic and non-diabetic patients in colonoscopy under sedoanalgesia | 24 hour
  After sedoanalgesia is applied respiratuar rate will be recorded.
Comparison of Ramsay sedation score level in diabetic and non-diabetic patients in colonoscopy under sedoanalgesia | 24 hour
  After sedoanalgesia is applied Ramsay sedation score level will be recorded. Ramsay sedation score level will be 3 during the process. When the score level is 2, at the end of the procedure, it will be taken to the postoperative intensive care unite.
Comparison of Modified post anaesthetic discharge score level in diabetic and non-diabetic patients in colonoscopy under sedoanalgesia | 24 hour
  After sedoanalgesia is applied modified post anaesthetic discharge score level will be recorded. Patients will be discharged when the score level is 9 or above.
Comparison of procedure times in diabetic and non-diabetic patients in colonoscopy under sedoanalgesia | 24 hour
  After sedoanalgesia is applied procedure times will be recorded.
Comparison of total anaesthetic doses in diabetic and non-diabetic patients in colonoscopy under sedoanalgesia | 24 hour
  After sedoanalgesia is applied total anaesthetic doses will be recorded.
Comparison of stomach ache and other effects in diabetic and non-diabetic patients in colonoscopy under sedoanalgesia | 24 hour
  After sedoanalgesia is applied stomach ache and other effects will be recorded. Stomach ache will be evaluated by visuel analog pain scale. When it is 4 or above, will be considered meaningful.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University Zubeyde Hanim Practice and Research Center, Izmir, Karşıyaka, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cho NH, Shaw JE, Karuranga S, Huang Y, da Rocha Fernandes JD, Ohlrogge AW, Malanda B. IDF Diabetes Atlas: Global estimates of diabetes prevalence for 2017 and projections for 2045. Diabetes Res Clin Pract. 2018 Apr;138:271-281. doi: 10.1016/j.diabres.2018.02.023. Epub 2018 Feb 26. PMID 29496507
- [Background] Zhao G, Ford ES, Ahluwalia IB, Li C, Mokdad AH. Prevalence and trends of receipt of cancer screenings among US women with diagnosed diabetes. J Gen Intern Med. 2009 Feb;24(2):270-5. doi: 10.1007/s11606-008-0858-8. Epub 2008 Dec 17. PMID 19089511
- [Background] Giovannucci E, Harlan DM, Archer MC, Bergenstal RM, Gapstur SM, Habel LA, Pollak M, Regensteiner JG, Yee D. Diabetes and cancer: a consensus report. Diabetes Care. 2010 Jul;33(7):1674-85. doi: 10.2337/dc10-0666. PMID 20587728
- [Background] Noto H, Tsujimoto T, Sasazuki T, Noda M. Significantly increased risk of cancer in patients with diabetes mellitus: a systematic review and meta-analysis. Endocr Pract. 2011 Jul-Aug;17(4):616-28. doi: 10.4158/EP10357.RA. PMID 21454235
- [Background] Yang X, Ko GT, So WY, Ma RC, Yu LW, Kong AP, Zhao H, Chow CC, Tong PC, Chan JC. Associations of hyperglycemia and insulin usage with the risk of cancer in type 2 diabetes: the Hong Kong diabetes registry. Diabetes. 2010 May;59(5):1254-60. doi: 10.2337/db09-1371. Epub 2010 Feb 25. PMID 20185812
- [Background] Renehan AG, Zwahlen M, Minder C, O'Dwyer ST, Shalet SM, Egger M. Insulin-like growth factor (IGF)-I, IGF binding protein-3, and cancer risk: systematic review and meta-regression analysis. Lancet. 2004 Apr 24;363(9418):1346-53. doi: 10.1016/S0140-6736(04)16044-3. PMID 15110491
- [Background] Diaz-Algorri Y, Lozada ME, Lopez SM, Bertran-Rodriguez CE, Gonzalez-Hernandez CM, Gonzalez D, Perez-Cardona CM, Hernandez J, Pedrosa C, Toro DH, Gonzalez-Pons M, Cruz-Correa M. Type 2 diabetes mellitus and colorectal neoplasia risk in Hispanics: a case-control study. J Diabetes Complications. 2015 May-Jun;29(4):502-7. doi: 10.1016/j.jdiacomp.2015.01.010. Epub 2015 Feb 3. PMID 25784088
- [Background] Vu HT, Ufere N, Yan Y, Wang JS, Early DS, Elwing JE. Diabetes mellitus increases risk for colorectal adenomas in younger patients. World J Gastroenterol. 2014 Jun 14;20(22):6946-52. doi: 10.3748/wjg.v20.i22.6946. PMID 24944487
- [Background] Kanadiya MK, Gohel TD, Sanaka MR, Thota PN, Shubrook JH Jr. Relationship between type-2 diabetes and use of metformin with risk of colorectal adenoma in an American population receiving colonoscopy. J Diabetes Complications. 2013 Sep-Oct;27(5):463-6. doi: 10.1016/j.jdiacomp.2013.04.010. Epub 2013 Jun 5. PMID 23755906
- [Background] Suh S, Kang M, Kim MY, Chung HS, Kim SK, Hur KY, Kim JH, Lee MS, Lee MK, Kim KW. Korean type 2 diabetes patients have multiple adenomatous polyps compared to non-diabetic controls. J Korean Med Sci. 2011 Sep;26(9):1196-200. doi: 10.3346/jkms.2011.26.9.1196. Epub 2011 Sep 1. PMID 21935276
- [Background] Giouleme O, Diamantidis MD, Katsaros MG. Is diabetes a causal agent for colorectal cancer? Pathophysiological and molecular mechanisms. World J Gastroenterol. 2011 Jan 28;17(4):444-8. doi: 10.3748/wjg.v17.i4.444. PMID 21274373
- [Background] Erbach M, Mehnert H, Schnell O. Diabetes and the risk for colorectal cancer. J Diabetes Complications. 2012 Jan-Feb;26(1):50-5. doi: 10.1016/j.jdiacomp.2011.11.003. Epub 2012 Feb 7. PMID 22321219
- [Background] Laish I, Mizrahi J, Naftali T, Konikoff FM. Diabetes Mellitus and Age are Risk Factors of Interval Colon Cancer: A Case-Control Study. Dig Dis. 2019;37(4):291-296. doi: 10.1159/000496740. Epub 2019 Feb 7. PMID 30731459
- [Background] Fanti L, Testoni PA. Sedation and analgesia in gastrointestinal endoscopy: what's new? World J Gastroenterol. 2010 May 28;16(20):2451-7. doi: 10.3748/wjg.v16.i20.2451. PMID 20503443
- [Background] Cornelius BW. Patients With Type 2 Diabetes: Anesthetic Management in the Ambulatory Setting. Part 1: Pathophysiology and Associated Disease States. Anesth Prog. 2016 Winter;63(4):208-215. doi: 10.2344/0003-3006-63.4.208. PMID 27973934
- [Background] Raz I, Hasdai D, Seltzer Z, Melmed RN. Effect of hyperglycemia on pain perception and on efficacy of morphine analgesia in rats. Diabetes. 1988 Sep;37(9):1253-9. doi: 10.2337/diab.37.9.1253. PMID 3410166
- [Background] Park SH, Bahk JH, Oh AY, Gil NS, Huh J, Lee JH. Gender difference and change of alpha(1)-adrenoceptors in the distal mesenteric arteries of streptozotocin-induced diabetic rats. Korean J Anesthesiol. 2011 Nov;61(5):419-27. doi: 10.4097/kjae.2011.61.5.419. Epub 2011 Nov 23. PMID 22148092
- [Background] Gul H, Yildiz O, Dogrul A, Yesilyurt O, Isimer A. The interaction between IL-1beta and morphine: possible mechanism of the deficiency of morphine-induced analgesia in diabetic mice. Pain. 2000 Dec 15;89(1):39-45. doi: 10.1016/S0304-3959(00)00343-2. PMID 11113291
- [Background] Karci A, Tasdogen A, Erkin Y, Aktas G, Elar Z. The analgesic effect of morphine on postoperative pain in diabetic patients. Acta Anaesthesiol Scand. 2004 May;48(5):619-24. doi: 10.1111/j.1399-6576.2004.00387.x. PMID 15101859
- [Background] deRoux SJ, Sgarlato A. Upper and lower gastrointestinal endoscopy mortality: the medical examiner's perspective. Forensic Sci Med Pathol. 2012 Mar;8(1):4-12. doi: 10.1007/s12024-011-9257-2. Epub 2011 Jun 11. PMID 21667169
- [Background] De Cosmo G, Congedo E, Lai C, Primieri P, Dottarelli A, Aceto P. Preoperative psychologic and demographic predictors of pain perception and tramadol consumption using intravenous patient-controlled analgesia. Clin J Pain. 2008 Jun;24(5):399-405. doi: 10.1097/AJP.0b013e3181671a08. PMID 18496304
- [Background] Uchiyama K, Kawai M, Tani M, Ueno M, Hama T, Yamaue H. Gender differences in postoperative pain after laparoscopic cholecystectomy. Surg Endosc. 2006 Mar;20(3):448-51. doi: 10.1007/s00464-005-0406-0. Epub 2006 Jan 21. PMID 16432649
- [Background] Mogil JS. Sex differences in pain and pain inhibition: multiple explanations of a controversial phenomenon. Nat Rev Neurosci. 2012 Dec;13(12):859-66. doi: 10.1038/nrn3360. PMID 23165262
- [Background] Newcomer MK, Shaw MJ, Williams DM, Jowell PS. Unplanned work absence following outpatient colonoscopy. J Clin Gastroenterol. 1999 Jul;29(1):76-8. doi: 10.1097/00004836-199907000-00019. PMID 10405238
- [Background] Takahashi Y, Tanaka H, Kinjo M, Sakumoto K. Prospective evaluation of factors predicting difficulty and pain during sedation-free colonoscopy. Dis Colon Rectum. 2005 Jun;48(6):1295-300. doi: 10.1007/s10350-004-0940-1. PMID 15793639
- [Background] Report of the Expert Committee on the Diagnosis and Classification of Diabetes Mellitus. Diabetes Care. 1997 Jul;20(7):1183-97. doi: 10.2337/diacare.20.7.1183. No abstract available. PMID 9203460
- [Background] Hochberg I, Segol O, Shental R, Shimoni P, Eldor R. Antihyperglycemic therapy during colonoscopy preparation: A review and suggestions for practical recommendations. United European Gastroenterol J. 2019 Jul;7(6):735-740. doi: 10.1177/2050640619846365. Epub 2019 Apr 20. PMID 31316777
- [Background] Ramsay MA, Savege TM, Simpson BR, Goodwin R. Controlled sedation with alphaxalone-alphadolone. Br Med J. 1974 Jun 22;2(5920):656-9. doi: 10.1136/bmj.2.5920.656. PMID 4835444
- [Background] Chung F, Chan VW, Ong D. A post-anesthetic discharge scoring system for home readiness after ambulatory surgery. J Clin Anesth. 1995 Sep;7(6):500-6. doi: 10.1016/0952-8180(95)00130-a. PMID 8534468
- [Background] Tuncali B, Pekcan YO, Celebi A, Zeyneloglu P. Addition of low-dose ketamine to midazolam-fentanyl-propofol-based sedation for colonoscopy: a randomized, double-blind, controlled trial. J Clin Anesth. 2015 Jun;27(4):301-6. doi: 10.1016/j.jclinane.2015.03.017. Epub 2015 Mar 20. PMID 25801162
- [Background] 31. Kayhan Z: Ağrının ölçülmesi: Klinik Anestezi 2019; Logos yayıncılık
- [Background] 32. Satman İ, Alagöl F, Ömer B, Kalaca S, Tütüncü Y, Çolak N. Türkiye Diyabet, Hipertansiyon, Obezite ve Endokrinolojik Hastalıklar Prevalans Çalışması-II. (TURDEP II) 2011.
- [Background] Joshi GP, Chung F, Vann MA, Ahmad S, Gan TJ, Goulson DT, Merrill DG, Twersky R; Society for Ambulatory Anesthesia. Society for Ambulatory Anesthesia consensus statement on perioperative blood glucose management in diabetic patients undergoing ambulatory surgery. Anesth Analg. 2010 Dec;111(6):1378-87. doi: 10.1213/ANE.0b013e3181f9c288. Epub 2010 Oct 1. PMID 20889933
- [Background] Cornelius BW. Patients With Type 2 Diabetes: Anesthetic Management in the Ambulatory Setting: Part 2: Pharmacology and Guidelines for Perioperative Management. Anesth Prog. 2017 Spring;64(1):39-44. doi: 10.2344/anpr-64-01-02. PMID 28128657